CLINICAL TRIAL: NCT05407298
Title: Prevalence of Cannabidiol (CBD) Consumption and Cancer Patients' Expectations in One Oncology Day-Hospital: A Cross-sectional Study and Questionnaire Validation
Brief Title: The Use of Cannabidiol in Cancer Patients
Acronym: CANPADIOL
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2022Ao001
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Cancer
Keywords: Cannabidiol; cancer patient
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CBD users
  Interventions: Other: Non applicable
- CBD non-users
  Interventions: Other: Non applicable

INTERVENTIONS:
Other: Non applicable — Non Applicable

SUMMARY:
Alternative and complementary medicines (MAC) are commonly used by cancer patients to help them to face with anticancer treatment, reduce oncology symptoms and/or anticancer treatment adverse effects, detoxifying the body. In consistence with guidelines from the French Society for Oncology Pharmacy (SFPO), the pharmaceutical consultation includes a discussion and collection of herbs, botanical and other natural products consumed by cancer patients. This aim to prevent and manage herb-drug interaction as well as other drug-related problems (DRP). The recent French experimentation dedicated to cannabidiol for medical use could enhance interest of cancer patients in the field of MAC. However, cannabidiol have shown inhibitory effect on different cytochromes with a risk of HDI as other MAC. While the prevalence of MAC consumption is already known in some type of cancer, the consumption of CBD is less known and should be explored. Through this study we wish to know the prevalence of cannabidiol consumption in cancer patients and to establish a typical profile as well as to know the modalities of use. We also want to validate a questionnaire through a literacy scale.

DETAILED DESCRIPTION:
* A Prospective observational study
* Conducted in an oncology day-hospital (CHU de Reims)

All data collected were:

* Clinical characteristics,
* Administrative data,
* Medication review,
* Biologic data collection,
* Oncological data,
* Disease data

Statistical analysis:

* Quantitative variables: described as mean ± standard deviation (SD) or median (Interquartile range and minimum and maximum)
* Student test and Fischer exact performed to compare CBD users and non-users.
* Analysis of variance: used to compare scores between different variables
* Univariate logistic and multivariate logistic regressions were performed. Variables with a p-value < 0.20 (Wald test) in the univariable analyses were considered eligible for the multivariable models.

ELIGIBILITY:
inclusion criteria: All the patients (>18yo) who received anticancer treatment

exclusion criteria:

* Patients who received anticancer drug with very short administration time (typically subcutaneous anticancer drugs as 5-azacitidine, bortezomib and some monoclonal antibodies)
* Patients who were not able to speak and understand French as well as who were unable to communicate clearly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients (>18yo) who received anticancer treatment during the inclusion period
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of CBD consummation among patients receiving anticancer treatment | Day 0

SECONDARY OUTCOMES:
Knowledge assessment of cancer patients with the CBD medical use in the literacy scope | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France